CLINICAL TRIAL: NCT06450314
Title: De-escalation of Medical Therapies in HER2-positive Metastatic Breast Cancer in Long-term Persistent Response and Minimal Residual Disease Undetectable in Circulating Tumor DNA
Brief Title: Decreasing Treatment for Metastatic HER2-Positive Breast Cancer With Undectable Cancer Levels in Blood Tests.
Acronym: HEROES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2312; 2023-509811-98-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer; HER2-positive Breast Cancer
Keywords: de-escalation; ctDNA test
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ctDNA negative cohort at baseline (Experimental): Patients with ctDNA negative test at baseline will stop their anti-HER2 targeted therapy during the study
  * In case of radiological progression with or without ctDNA positive test, prior treatment will be restarted or new anti-HER2 treatment will be initiated according investigator choice
  * In case of ctDNA positive test without radiological progression, prior treatment will be restarted.
  Interventions: Drug: Discontinuation of the anti-HER2 maintenance therapy; Device: Monitoring with signatera test

INTERVENTIONS:
Drug: Discontinuation of the anti-HER2 maintenance therapy — Heroes is a de-escalation study. Patient must have received continuous anti-HER2 targeted therapy (including Trastuzumab, Trastuzumab/Pertuzumab, Trastuzumab-Deruxtecan, T-DM1) for at least 2 years in any line setting for their HER2-positive metastatic breast cancer with complete response or partial response at last radiological assessment. Patients with ctDNA negative test at baseline will stop their anti-HER2 targeted therapy during the study
Device: Monitoring with signatera test — ctDNA test will be performed at 1.5 month after inclusion and every 3 months during 2 years.
  Note: For the ctDNA negative patients who become ctDNA positive: ctDNA test will be performed once, 3 months after restarting treatment (+/-1 week).

SUMMARY:
Heroes is a multicentre, national, non-randomized, open-label, phase 2 study. The goal of this clinical trial is to evaluate the feasibility of therapeutic de-escalation in HER2-positive metastatic breast cancer with disease controlled after 2 years of maintenance treatment with anti-HER2 targeted therapy AND ctDNA negative testing.

The main question it aims to answer is :

• Is it possible to identify patients for whom temporary or permanent discontinuation of treatment is possible without impacting prognosis?

DETAILED DESCRIPTION:
Metastatic breast cancer remains a difficult disease to cure in the majority of cases. Improved biological knowledge has made it possible to separate these heterogeneous pathologies into several subtypes. For the HER2 subtype, which accounts for around 15% of breast cancers, very significant progress has been made in recent years with innovative treatments known as anti-HER2 therapies (trastuzumab, pertuzumab, T-DM1, T-DXd). Long-term disease control has been achieved in at least 20% of these patients with these new treatments.

However, the treatments are continued indefinitely, impacting patients' quality of life through toxicity and chronic administration. It is possible that, for some patients, these treatments can be discontinued while maintaining surveillance. To assess this possibility, new biological tools, notably the search for circulating tumor DNA (ctDNA), look very promising for detecting any tumor cells in the body, even to very small traces (minimal residual disease).

The primary objective of this trial is to evaluate the feasibility of therapeutic de-escalation (temporary or complete discontinuation) in patients with HER2-positive metastatic breast cancer whose disease is controlled after 2 years of maintenance treatment with anti-HER2 targeted therapy AND a negative ctDNA test.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in signing the patient's consent;
2. Men or women ≥18 years of age;
3. Documented diagnosis of locally advanced inoperable or metastatic histologically-proven HER2-positive breast cancer (HER2-positive is defined as HER2 3+ immunohistochemical overexpression, or the presence of HER2 amplification, according to ASCO-CAP guidelines);
4. Must have an adequate archival tumor tissue sample available for next-generation sequencing (NGS) analysis by central laboratory, in order to design the ctDNA test (based on most recent available tumor tissue sample, metastatic biopsy (bone tissue excluded) and primary tumor authorised);
5. Patient with Eastern Cooperative Oncology Group - Performance Status (ECOG-PS) ≤1;
6. Patient must have received continuous anti-HER2 targeted therapy (including Trastuzumab, Trastuzumab/Pertuzumab, Trastuzumab-Deruxtecan or T-DM1) treatment for at least 2 years in any line setting, for their locally advanced inoperable or metastatic HER2 + breast cancer (prior treatment interruption of 3 months maximum is allowed), with complete response or partial response at last radiological assessment;

   Note: the number of patients who received anti-HER2 targeted therapy in second line setting or more will be capped to 50% of the overall population
7. In case of bone disease only, complete metabolic response in 18-FDG pet-scanner is required;
8. Patient with treated (surgery and/or radiation therapy) and controlled primary tumor;
9. Patients with ER-positive disease may or may not have received concomitant endocrine therapy (which must be continued if present). Concomitant ovarian blockade using Luteinizing Hormone-Releasing Hormone (LHRH) agonists is authorised as well;
10. Adequate cardiac, renal, haematological and hepatic functions according to guidelines hospital;
11. Women of childbearing potential must have a negative serum or urine pregnancy test done within 28 days before inclusion;
12. Non post-menopausal women and fertile men must agree to use adequate contraception methods during the study. Hormonal contraceptives such as birth control pills, patches, implants, or injections are not allowed in patients who are hormone receptor positive;
13. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan and other study procedures including follow-up;
14. Patients must be affiliated to a Social Security System (or equivalent).

Exclusion Criteria:

1. Any breast cancer progression over the past 2 years or at study entry;
2. Patient concurrently using other approved or investigational antineoplastic agents than trastuzumab, pertuzumab, Trastuzumab-Deruxtecan, TDM-1 +/- endocrine therapy;
3. Had an history of tumoral meningitis or clinically active central nervous system metastases, defined as untreated or symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms;

   1. Subjects with curatively treated brain metastases (i.e., complete removal surgery or stereotactic radiotherapy) who are no longer symptomatic and do not require treatment with corticosteroids or anticonvulsants may be included in the study provided they have recovered from the acute toxicity of radiotherapy and there has been no progression of the brain metastases within the past 24 months.
   2. Subjects with brain metastases only or treated with whole brain radiotherapy will be excluded of the study
4. Major concurrent disease affecting cardiovascular system, liver, kidneys, haematopoietic system or else considered as clinically important by the investigator and that could be incompatible with patient's participation in this trial or would likely interfere with study procedures or results;
5. History of any prior ipsi or contralateral breast cancer (except in case of DCIS) unless if both primary tumors were confirmed to be HER2-positive;
6. Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease and treatment for at least 3 years;
7. Major surgery within 2 weeks prior to study entry;
8. Pregnant women or women who are breast-feeding;
9. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons;
10. Participation in another clinical study whose procedures interfere with those of the study (within 28 days prior to patient enrolment and for the duration of the study);
11. Persons deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free rate | 1 year
  The progression-free rate (PFR) is the percentage of patient with disease progression defined as the time from the date of registration to the date of the first documented event among radiological progressions (RECIST 1.1), molecular progressions definitive as ctDNA-positive results, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival | 1 year
  Progression-free survival (PFS) is defined as the time from the date of registration to the date of the first documented cancer progression measured by RECIST 1.1 or death due to any cause, whichever occurs first.
ctDNA dynamics | 1 year
  The ctDNA dynamics is defined as changes in the level of ctDNA (from negative to positive) during the surveillance phase.
ctDNA positivity rate | 1 year
  Positivity rate is defined as the proportion of patients with positive ctDNA results.
Overall Survival | 1 year
  Overall Survival (OS) is defined as the time from the date of registration to the date of death due to any cause
Molecular response | 1 year
  Molecular response is defined as the percentage of patients who reached molecular remission (ctDNA clearance) 3 months after reintroduction of anti-HER2 treatment among patients with ctDNA positive without RECIST progression.
Objective Response Rate | 1 year
  Objective Response Rate (ORR) is defined as the number of patients with at least a confirmed complete response (CR) or partial response (PR) to reintroduction of anti-HER2 treatment, among patients with RECIST progression during the surveillance phase
Duration of Response | 1 year
  The duration of response (Dor) is defined, among patients with RECIST progression during the surveillance phase, as the time from the onset of response after reintroduction of anti-HER2 treatment, to progression or death due to any cause, whichever occurs first.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline then every 3 months during 2 years and every 6 months the third year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Breast cancer module (QLQ-BR45) | At baseline then every 3 months during 2 years and every 6 months the third year
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR45 incorporates nine multi-item scales to assess body image, sexual functioning, breast satisfaction, systemic therapy side effects, arm symptoms, breast symptoms, endocrine therapy symptoms, skin mucosis symptoms, endocrine sexual symptoms. In addition, single items assess sexual enjoyment, future perspective and being upset by hair loss. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. Higher scores indicate more severe symptoms or problems.
State-Trait Anxiety Inventory - state (STAI-S) | At 6 months and 1 year
  The State-Trait Anxiety Inventory - state (STAI-S) is a commonly used measure of state anxiety.
  This 20-item questionnaire measures the intensity of the participant's anxiety at the moment of testing. The items are designed to measure an individual's feelings oftension, apprehension, nervousness, and worry. All items are rated on a 4-point scale (1 = "not at all", 2 = "somewhat", 3 = "moderately", and 4 = "very much"). Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Decision regret scale (DRS) | At 6 months and 1 year
  The decision regret was developed to measure regret after health-care decisions.
  This questionnaire incorparate 5 items about decision regret, decision correctness, belief in making the same decision again, wisdom and any resulting harm from the decision. All items are rated on a 5-point Likert-type scale (1 = "strongly agree", 2 = "agree", 3 = "neither agree or disagree", 4 = "disagree", and 5 = "strongly disagree"), and are transformed to a 0-100 scale. Higher scores indicate more regret.

CONTACTS AND LOCATIONS:
Overall Officials: Thibault De la Motte Rouge, MD, Principal Investigator — Centre Eugene Marquis
Locations (1):
- Centre Eugène marquis, Rennes, France

IPD SHARING:
Plan to Share IPD: No